CLINICAL TRIAL: NCT04495010
Title: A Phase 2, Randomized Study of Neoadjuvant Nivolumab Plus Ipilimumab Followed by Adjuvant Nivolumab or Neoadjuvant Nivolumab Plus Ipilimumab Followed by Either Adjuvant Nivolumab or Postsurgical Observation Depending on Pathologic Response Compared With Adjuvant Nivolumab in Treatment-Naive Patients With Resectable Clinically Detectable Stage III Melanoma
Brief Title: Neoadjuvant Nivolumab+Ipilimumab Followed by Adjuvant Nivolumab or Neoadjuvant Nivolumab+Ipilimumab Followed by Adjuvant Observation Compared With Adjuvant Nivolumab in Treatment-Naive High-risk Melanoma Participants
Acronym: CheckMate 7UA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-7UA; 2020-000070-16 (EudraCT Number)
Record Dates: First submitted 2020-07-30; First posted 2020-07-31 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Neoadjuvant treatment + Adjuvant treatment (Experimental)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Adjuvant treatment (Experimental)
  Interventions: Biological: Nivolumab
- Neo treat with patho response-driven Adju treat or observation (Experimental): Neoadjuvant treatment with pathologic response-driven Adjuvant treatment or observation
  Interventions: Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo
Biological: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy
  Arms: Neo treat with patho response-driven Adju treat or observation; Neoadjuvant treatment + Adjuvant treatment

SUMMARY:
The purpose of this study is to evaluate the role of neoadjuvant immunotherapy and to demonstrate high pathologic complete response (pCR) and near pCR rates in melanoma participants with clinically detectable nodal disease and a high risk of recurrence. Neoadjuvant immunotherapy aims to enhance the systemic T-cell response to tumor antigens while detectable tumor is still present, inducing a stronger and broader tumor-specific immune response. Of the neoadjuvant approaches studied within melanoma, the neoadjuvant combination of nivolumab and ipilimumab has demonstrated high pCR and near pCR rates that may translate to prolonged clinical benefit.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Males and females, ≥ 12 years of age [Except: where local regulations and/or institutional policies do not allow for participants < 18 years of age (adolescent population) to participate. For those sites, the eligible participant population is 18 years of age or local age of majority, inclusive]
* Diagnosed with cytologically or histologically confirmed Stage IIIB, IIIC, or IIID cutaneous melanoma as per American Joint Committee on Cancer (AJCC) staging system, with ≥ 1 clinically detectable lymph node metastases (N1b, N2b, N3b), which are measurable according to Response Evaluation Criteria In Solid Tumors version 1.1 (RECIST 1.1)
* Adult participants and adolescents 16 to 18 years old must have an Eastern Cooperative Oncology Group (ECOG) scale performance status of 0 or 1. Adolescents < 16 years old must have Lanksky Play-Performance Status scale performance of ≥ 60
* Must be treatment-naïve (ie, no prior systemic anticancer therapy as adjuvant therapy for melanoma or unresectable/metastatic melanoma)
* Women and men must agree to follow specific methods of contraception, if applicable, while participating in the trial

Exclusion Criteria:

* Women who are breastfeeding
* Patients with serious or uncontrolled medical disorders
* Prior treatment with an anti-programmed cell death protein 1 (PD-1), anti-programmed death-ligand 1 (PD-L1), anti-programmed death-ligand 2 (PD-L2), or anti cytotoxic T-lymphocyte antigen 4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-31 (Estimated); Primary Completion 2024-02-28 (Estimated); Study Completion 2027-10-23 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | Up to 4 years

SECONDARY OUTCOMES:
Recurrence-free survival (RFS) Time from Surgery | Up to 5 years
RFS Time from Adjuvant Therapy | Up to 5 years
Pathologic response rate (pRR) by immune-related pathologic response (irPR) | Up to 5 years
Concordance major pathologic response (MPR) by local and central pathology Review | Up to 5 years
  MPR is defined as participants achieving either pathologic complete response (pCR) or near pCR
RFS by MPR | Up to 5 years
Incidence of Adverse Events (AEs) | Up to 5 years
Incidence of Serious Adverse Events (SAEs) | Up to 5 years
Incidence of deaths | Up to 5 years
Incidence of clinically significant changes in clinical laboratory results: Hematology tests | Up to 5 years
Incidence of clinically significant changes in clinical laboratory results: Clinical Chemistry tests | Up to 5 years
Incidence of clinically significant changes in clinical laboratory results: Urinalysis tests | Up to 5 years
Change from baseline in Health-related quality of life (HRQoL) by the Trial Outcome Index (TOI) and Melanoma Subscale (MS) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (108):
- United States (20):
  - Local Institution, Gilbert, Arizona
  - Local Institution, Tucson, Arizona
  - Local Institution, San Francisco, California
  - Local Institution, Aurora, Colorado
  - Local Institution, Tampa, Florida
  - Local Institution, Atlanta, Georgia
  - Local Institution, Marietta, Georgia
  - Local Institution, Annapolis, Maryland
  - Local Institution, Boston, Massachusetts
  - Local Institution, Minneapolis, Minnesota
  - Local Institution, Hattiesburg, Mississippi
  - Local Institution, St Louis, Missouri
  - Local Institution, Morristown, New Jersey
  - Local Institution, New Brunswick, New Jersey
  - Local Institution, Cleveland, Ohio
  - Local Institution, Portland, Oregon
  - Local Institution, Houston, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Charlottesville, Virginia
  - Local Institution, Seattle, Washington
- Australia (10):
  - Local Institution, North Sydney, New South Wales
  - Local Institution, Westmead, New South Wales
  - Local Institution, Greenslopes, Queensland
  - Local Institution, Woolloongabba, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Hobart, Tasmania
  - Local Institution, Ballarat, Victoria
  - Local Institution, Melbourne, Victoria
  - Local Institution, Doubleview, Western Australia
  - Local Institution, Nedlands, Western Australia
- Austria (5):
  - Local Institution, Graz
  - Local Institution, Innsbruck
  - Local Institution, Salzburg
  - Local Institution, Sankt Pölten
  - Local Institution, Vienna
- Belgium (3):
  - Local Institution, Brussels
  - Local Institution, Ghent
  - Local Institution, Wilrijk
- Brazil (8):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Brasília, Federal District
  - Local Institution, Curitiba, Paraná
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Florianópolis, Santa Catarina
  - Local Institution, São José do Rio Preto, São Paulo
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Denmark (3):
  - Local Institution, Aarhus
  - Local Institution, Herlev
  - Local Institution, Odense C
- France (12):
  - Local Institution, Bordeaux
  - Local Institution, Dijon
  - Local Institution, Lille
  - Local Institution, Marseille
  - Local Institution, Nantes
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Pierre-Bénite
  - Local Institution, Rennes
  - Local Institution, Sr Priest En Jarez
  - Local Institution, Toulouse
  - Local Institution, Villejuif
- Germany (11):
  - Local Institution, Berlin
  - Local Institution, Erlangen
  - Local Institution, Essen
  - Local Institution, Hanover
  - Local Institution, Heidelberg
  - Local Institution, Kiel
  - Local Institution, Lübeck
  - Local Institution, Mainz
  - Local Institution, Regensburg
  - Local Institution, Tübingen
  - Local Institution, Würzburg
- Italy (6):
  - Local Institution, Bergamo
  - Local Institution, Meldola
  - Local Institution, Napoli
  - Local Institution, Novara
  - Local Institution, Padua
  - Local Institution, Pavia
- Netherlands (6):
  - Local Institution, Amsterdam
  - Local Institution, Breda
  - Local Institution, Geleen
  - Local Institution, Leiden
  - Local Institution, Rotterdam
  - Local Institution, Utrecht
- Poland (3):
  - Local Institution, Krakow
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
- Russia (3):
  - Local Institution, Krasnodar
  - Local Institution, Ryazan
  - Local Institution, Saint Petersburg
- Spain (7):
  - Local Institution, Barcelona
  - Local Institution, Haddon Heights
  - Local Institution, Madrid
  - Local Institution, Málaga
  - Local Institution, Oviedo
  - Local Institution, Santiago de Compostela
  - Local Institution, Seville
- Local Institution, Vaxjo, Sweden
- Local Institution, Zurich, Switzerland
- United Kingdom (9):
  - Local Institution, Cambridge
  - Local Institution, Glasgow
  - Local Institution, Guildford
  - Local Institution, Leeds
  - Local Institution, London
  - Local Institution, Manchester
  - Local Institution, Northwood
  - Local Institution, Oxford
  - Local Institution, Sutton

REFERENCES:
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm